CLINICAL TRIAL: NCT05227456
Title: Failed Endometrial Ablation Treatment With Implantable Progesterone (FEAT) Study
Acronym: FEATS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in Recruitment
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Sarah Smith, Obstetrician Gynecologist, Principal Investigator, Assistant Professor, Saskatchewan Health Authority - Regina Area
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB-22-05
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Abnormal Uterine Bleeding; Dysmenorrhea
Keywords: abnormal uterine bleeding; pain; dysmenorrhea; endometrial ablation
MeSH Terms: conditions — Metrorrhagia; Dysmenorrhea; Pain | interventions — etonogestrel; Drug Implants; Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Etonogestrel implant (Experimental): The participants will receive an etonogestrel 68mg implant
  Interventions: Drug: Etonogestrel 68mg implant; Device: Etonogestrel 68mg implant

INTERVENTIONS:
Drug: Etonogestrel 68mg implant — Implant will be inserted
  Other Names: Nexplanon
Device: Etonogestrel 68mg implant — Implant will be inserted
  Other Names: Nexplanon

SUMMARY:
The objective of this study is to assess the efficacy of an implantable etonogestrel device in reducing hysterectomy rate in patients with a failed endometrial ablation.

DETAILED DESCRIPTION:
The researchers aim to determine whether use of etonogestrel implant in patients with failed endometrial ablation significantly decreases hysterectomy rate. Changes in pelvic pain and vaginal bleeding will be assessed. Time to hysterectomy will be examined.

The researchers hypothesize that treatment of failed endometrial ablation with etonogestrel implant will decrease pelvic pain and vaginal bleeding resulting in a significantly decreased need for hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Previous endometrial ablation
* Pelvic pain and/or vaginal bleeding seeking treatment

Exclusion Criteria:

* Previous or current VTE
* Liver tumour, benign or malignant, or active liver disease
* Undiagnosed abnormal genital bleeding
* Known or suspected breast cancer
* Uncontrolled hypertension
* Allergy to component of etonogestrel implant
* Lack of patient consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Hysterectomy | Occurrence of hysterectomy will be documented any time during the 3 year follow up period
  occurrence of hysterectomy

SECONDARY OUTCOMES:
Vaginal bleeding | PBAC score will be documented at baseline and 3, 6, 12, 18, 24, 30, and 36 months
  Pictorial Blood Loss Assessment Chart (PBAC) score, minimum score = 0mL, maximum score = n/a, higher score indicates higher menstrual blood loss
Pelvic Pain | VAS will be documented at baseline and 3, 6, 12, 18, 24, 30, and 36 months
  Assessment of pelvic pain using Visual Analogue Scale (VAS), minimum score = 0, maximum score = 10, higher score indicates more pain
Time to Hysterectomy | Time of hysterectomy will be documented any time during the 3 year follow up period
  Time from booking of hysterectomy to actual hysterectomy will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Sarah N Smith, MD, Principal Investigator — Obstetrician Gynecologist
Locations (1):
- Saskatchewan Health Authority, Regina, Saskatchewan, Canada